CLINICAL TRIAL: NCT01160588
Title: Brain Markers of Anxiety Disorders and SSRI/CBT Treatment in Children and Adolescents
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, K. Luan Phan, Principal Investigator; Associate Professor, University of Michigan
Other Study IDs: R01MH086517 (NIH); R01MH086517 (NIH)
Record Dates: First submitted 2010-07-09; First posted 2010-07-12 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Social Phobia; Generalized Anxiety Disorder; Separation Anxiety Disorder
Keywords: Anxiety; Social Phobia; Social Anxiety; Generalized Anxiety; Separation Anxiety
MeSH Terms: conditions — Phobia, Social; Generalized Anxiety Disorder; Anxiety, Separation; Anxiety Disorders | interventions — Sertraline

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — saliva
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Sertraline treatment: Participants with Generalized Anxiety Disorder, and/or Social Anxiety Disorder, and/or Separation Anxiety Disorder will undergo MRI scanning, EEG's, and sertraline treatment.
  Interventions: Drug: Sertraline
- Healthy Controls: Healthy control participants will undergo MRI scanning and EEG's.
- Cognitive Behavioral Therapy: Participants with Generalized Anxiety Disorder, and/or Social Anxiety Disorder, and/or Separation Anxiety Disorder will undergo MRI scanning, EEG's, and talk therapy (CBT).

INTERVENTIONS:
Drug: Sertraline — Oral sertraline will be started at 25 mg/day, increasing on subsequent visits to 50, 75, 100, 125, 150, and 200mg/day) Unless adverse effects become problematic, the goal is for subjects to reach 200mg/day. Dosing of sertraline is flexible, based on tolerance (absence of side effects) and clinical response.
  Other Names: Zoloft
  Groups: Sertraline treatment

SUMMARY:
This study will attempt to identify gene and brain activity markers that predict whether children and adolescents with anxiety disorders will respond to selective serotonin reuptake inhibitor medications or Cognitive Behavioral Therapy (CBT).

DETAILED DESCRIPTION:
Anxiety disorders are common and highly disabling conditions of children and adolescence that often do not remit, and increase the risk of depression, anxiety, substance abuse, and suicide in adulthood. Available treatments are only modestly successful. When they are effective, however, early treatment of anxiety disorders can reduce subsequent morbidity.

This study will examine variations in genetics and brain reactivity among children and adolescents who do and do not respond to SSRIs and Cognitive Behavioral Therapy. Through this, the study will identify neurological and genetic biomarkers that can predict responsiveness to SSRI/CBT treatment in those with anxiety disorders.

For SSRI/medication treatment arm:

Although selective serotonin reuptake inhibitors (SSRI) are medications widely prescribed for children and adolescents with anxiety disorders, little is known about the neurobiological factors that predict which patients respond to treatment. Current theory suggests that neurological functioning and genetics may influence a patient's response to treatment.

Participation in this study will last approximately 14 weeks. Both healthy participants and participants with anxiety disorders will be recruited to participate. All participants will complete similar study visits at entry, within 2 weeks of entry, and 12 weeks after that. The first visit, which will occur at study entry, will include screening questionnaires, an interview with research staff, a medical screening, and collection of saliva samples for genotyping. The second visit and the last visit, which will be separated by 12 weeks, will involve MRI scans and behavioral tasks to be conducted inside and outside the MRI scanner. Over the 12 weeks between MRI scanning sessions, participants with anxiety disorders will take sertraline, a common SSRI, on a daily basis. They will also attend nine additional visits during this time to complete assessments of their symptoms. These visits will occur 0, 1, 2, 3, 4, 6, 8, 10 and 12 weeks after the first scan. Participants with anxiety disorders will therefore be completing a symptom assessment, MRI scans, and behavioral tasks all on the final visit, 12 weeks after the second visit. In addition, participants will complete tasks while connected to an Electroencephalography(EEG) machine before and after the 12 weeks of treatment, and will have the option of additional EEG's at weeks 2, 4, and 8.

For CBT arm:

Participation in this study will last 16 weeks. All participants will complete similar study visits at entry, within 2 weeks of entry, and approximately 16 weeks after that. The first visit, which will occur at study entry, will include screening questionnaires, an interview with research staff, a medical screening, and collection of saliva samples for genotyping. The second visit and the last visit, which will be separated by approximately 16 weeks, will involve MRI scans and behavioral tasks to be conducted inside and outside the MRI scanner. Over the 16 weeks between MRI scanning sessions, participants with anxiety disorders will participate in type of talk therapy--Cognitive Behavioral Therapy--on a weekly basis. In addition, participants will complete tasks while connected to an Electroencephalography(EEG)machine before and after the 16 weeks of treatment, and will have the option of additional EEG's at weeks 2, 4, and 8.

ELIGIBILITY:
Inclusion Criteria:

For anxiety disorder group:

* 7-19 years of age
* Current diagnosis of social anxiety disorder, generalized anxiety disorder and/or separation anxiety disorder
* Physically healthy, as confirmed by comprehensive medical history, physical exam, and laboratory testing

For healthy control group:

* 7-19 years of age
* Never been diagnosed with either Axis I or Axis II mental disorders
* Physically healthy, as confirmed by comprehensive medical history, physical exam, and laboratory testing

Exclusion Criteria for all:

* Clinically significant medical or neurologic condition
* Life history of bipolar disorder, schizophrenia, mental retardation, or pervasive developmental disorder or current alcohol/drug abuse or dependence
* Severe current depression, as indicated by the Child Depression Inventory, or by the clinical decision of the rater or doctor
* Current suicidal ideation
* Treatment with psychotropic/psychoactive medications in the past two weeks (4 weeks for fluoxetine and monoamine oxidase inhibitors) before screening
* Positive urine drug screen results
* Pregnancy
* Clinically significant medical condition that interferes with metabolism of sertraline
* Multiple drug allergies
* Prior failure of response to sertraline for anxiety, as defined by adequate duration to achieve a clinical response
* Refusing to attend school because of anxiety

Additional exclusion criteria for the functional MRI studies:

* Presence of ferrous-containing metals within the body, such as aneurysm clips, shrapnel, or retained particles
* Claustrophobia

Ages: 7 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Participants with one or more of the following anxiety disorders (diagnosed by our study): Generalized Anxiety Disorder, Social Anxiety Disorder, Separation Anxiety Disorder.
Sampling Method: Non-Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2010-07; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Clinical Global Impression (CGI) Scale | Change from Baseline in CGI score at 12 or 16 weeks after treatment SSRI or CBT, respectively). Measured before treatment, at each treatment study visits, and after treatment

SECONDARY OUTCOMES:
Liebowitz Social Anxiety Scale (LSAS) | Change from Baseline in LSAS score at 12 or 16 weeks after treatment SSRI or CBT, respectively). Measured before treatment, at each treatment study visits, and after treatment

CONTACTS AND LOCATIONS:
Overall Officials: K. Luan Phan, M.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States